CLINICAL TRIAL: NCT02377895
Title: A Single-Center, Double-Masked, Randomized, Placebo-Controlled, Parallel-Group Allergen BioCube Study Evaluating the Efficacy and Safety of Nasapaque Nasal Solution in a Population of Adult Subjects With Seasonal Allergic Rhinitis
Brief Title: Allergen Biocube Study Evaluating Efficacy and Safety of Nasapaque Nasal Solution in Adult Subjects With Allergic Rhinitis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: 3E Therapeutics Corporation (Industry)
Collaborators: ORA, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 14-100-0008
Record Dates: First submitted 2015-02-27; First posted 2015-03-04 (Estimated); Last update posted 2017-01-26 (Estimated); Status verified 2017-01

CONDITIONS: Seasonal Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nasapaque Nasal Solution (Experimental): 250 ul in each nostril at Day 1 and Day 8
  Interventions: Drug: Nasapaque Nasal Solution
- Placebo Saline Nasal Solution (Active Comparator): 250 ul in each nostril at Day 1 and Day 8
  Interventions: Drug: Placebo Saline Nasal Solution

INTERVENTIONS:
Drug: Nasapaque Nasal Solution
  Arms: Nasapaque Nasal Solution
Drug: Placebo Saline Nasal Solution
  Arms: Placebo Saline Nasal Solution

SUMMARY:
Single-center, double-masked, randomized, placebo-controlled, parallel-group, efficacy and safety study using the Allergen BioCube (ABC).

ELIGIBILITY:
Key Inclusion Criteria:

* Must be 18 years of age and provide written informed consent and sign the HIPAA form
* Must have history of allergic rhinitis
* Must have positive response to Allergen BioCube

Key Exclusion Criteria:

* Must not have a significant illness such as moderate to severe allergic asthmatic reactions
* Must not have compromised lung function
* Must not use any disallowed medications
* Must not have been in an investigational study in the last 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2015-03; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
TNSS Total Nasal Symptom Score | Day 1 and Day 8

SECONDARY OUTCOMES:
Nasal Inspiratory Flow | Day 1 and Day 8
Nasal Inflammation Score | Day 1 and Day 8

REFERENCES:
- [Derived] Gomes PJ, Abelson MB, Stein L, Viirre E, Villafranca JE, Lasser EC. Iodixanol nasal solution reduces allergic rhinoconjunctivitis signs and symptoms in Allergen BioCube(R): a randomized clinical trial. J Asthma Allergy. 2019 Mar 1;12:71-81. doi: 10.2147/JAA.S150251. eCollection 2019. PMID 30881050